CLINICAL TRIAL: NCT02397408
Title: Phase 2 Study of 11C- and 18F-Choline PET/MR Imaging in Patients With Unfavorable Intermediate to High-Risk Prostate Cancer
Brief Title: 11C- and 18F-Choline PET/MR Imaging for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Albert J. Chang, MD, PhD, Assistant Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 145511; NCI-2015-00731 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); R01CA148708 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-03-25 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluorocholine; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic 11C- and 18F-choline PET/MR imaging (Experimental): Patients are given 370 megabecquerel (MBq) 11C-Choline (11C) intravenously and 3 MBq/kg 18F-Choline (18F) intravenously prior to a whole-body PET/MR imaging
  Interventions: Drug: Carbon C 11 Choline; Drug: Fluorine F 18 Choline; Procedure: Positron Emission Tomography (PET) / Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: Carbon C 11 Choline — Given intravenously (IV) prior to imaging
  Other Names: C-11 Choline; Ethanaminium, 2-hydroxy-N,N-dimethyl-N-(methyl-11C)-
Drug: Fluorine F 18 Choline — Given intravenously (IV) prior to imaging
  Other Names: 18F-Fluorocholine; [18F]-Choline
Procedure: Positron Emission Tomography (PET) / Magnetic Resonance Imaging (MRI) — Undergo whole-body PET/MR imaging
  Other Names: PET/MRI; Whole-body PET/MR imaging

SUMMARY:
This phase II trial studies how well 11C-choline (carbon C 11 choline) and 18F-choline (fluorine F 18 choline) positron emission tomography/magnetic resonance (PET/MR) imaging works in diagnosing patients with unfavorable intermediate to high-risk prostate cancer. Diagnostic procedures, such as 11C- and 18F-choline PET/MR may help find and diagnose prostate cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the ability of 11C- and 18F-choline PET/MR to detect and localize prostate cancer within the prostate gland.

SECONDARY OBJECTIVES:

I. To assess the ability of 11C- and 18F-choline PET/MR to detect the specific location of metastatic prostate cancer within pelvic lymph node regions in patients undergoing radical prostatectomy and extended pelvic lymph node dissection.

II. To assess the comparative performance of 11C- and 18F-choline PET/MR to already available imaging scans (bone scan, sodium fluoride positron emission tomography/computed tomography [NaF PET/CT], multiparametric1H magnetic resonance imaging [MRI], and/or pelvic CT scans) for detecting and localization of disease within the prostate, lymph nodes, and distant metastatic sites.

III. To determine the temporal distribution of 11C- and 18F-choline radiotracer in patients. The tissue uptake, retention, and clearance will be determined.

EXPLORATORY OBJECTIVES:

I. To compare regions of uptake on the 11C- and 18F-choline PET/MR to that on the sentinel lymph node imaging scans in patients undergoing sentinel lymph node-guided extended pelvic lymph node dissection.

OUTLINE:

Patients undergo 11C- and 18F-choline whole-body PET/MR imaging. After completion of study treatment, patients are followed up for 3 hours

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be >=18 years of age
* Diagnosis: Patients must have a diagnosis of prostate cancer by histologic verification and a hypoechoic lesion seen on ultrasound.
* Disease Status: Unfavorable intermediate to high-risk prostate cancer, per the Cancer of the Prostate Risk Assessment Score (CAPRA) (CAPRA 5-10)
* Karnofsky Performance Status >=70
* Metastatic workup: Whole Body Sodium Fluoride (NaF) PET/CT or 99mTc Bone Scan
* Planned to undergo radical prostatectomy and extended pelvic lymph node dissection
* Adequate bone marrow and organ function defined as follows:
* Adequate bone marrow function:
* Leukocytes >= 3,000/microliter (mcL)
* Absolute Neutrophil Count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Adequate hepatic function:
* Total bilirubin - within normal institutional limits
* Aspartate aminotransferase (AST)/ serum glutamic-oxaloacetic transaminase (SGOT) <= 2.5 X institutional upper limit of normal
* Alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) <= 2.5 X institutional upper limit of normal
* Adequate renal function:
* Creatinine - within normal institutional limits OR
* Creatinine clearance >= 60 mL/min/ 1.73m2 for patients with creatinine levels above institutional normal
* Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

* Participation would significantly delay the scheduled standard of care therapy
* Karnofsky performance status of < 60
* Inadequate venous access
* Administered a radioisotope within 5 physical half lives prior to study enrollment
* Have a medical condition or other circumstances which, in the opinion of the investigator would significantly decrease the chances of obtaining reliable data, achieving the study objectives, or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-04-09 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert J Chang, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choi JY, Yang J, Noworolski SM, Behr S, Chang AJ, Simko JP, Nguyen HG, Carroll PR, Kurhanewicz J, Seo Y. 18F Fluorocholine Dynamic Time-of-Flight PET/MR Imaging in Patients with Newly Diagnosed Intermediate- to High-Risk Prostate Cancer: Initial Clinical-Pathologic Comparisons. Radiology. 2017 Feb;282(2):429-436. doi: 10.1148/radiol.2016160220. Epub 2016 Aug 11. PMID 27513849
- See also: Link to Publication for NCT02397408 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5283870/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Division of Radiation Oncology, Division Urological Medical Oncology, and the Division of Urologic Surgical Oncology at the Helen Diller Family Comprehensive Cancer Center at University of California, San Francisco (UCSF) who are planning to undergo radical prostatectomy of definitive radiation therapy.
Groups:
- Diagnostic 11C- and 18F-choline PET/MR Imaging: Patients are given 370MBq 11C-Choline intravenously and 3MBq/kg 18F-Choline intravenously prior to a whole-body PET/MR imaging
Period: Overall Study
Arm/Group | Diagnostic 11C- and 18F-choline PET/MR Imaging
Started | 18
Completed Surgery Per Protocol | 16
Completed | 12
Not Completed | 6
Not completed — Physician Decision | 4
Not completed — Surgery not completed within protocol timeframe | 2

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic 11C- and 18F-choline PET/MR Imaging
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 5
  60-69 years old | 8
  70-79 years old | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 18
Serum Prostate-Specific Antigen (PSA) Level [Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)] — Prostate-specific antigen (PSA) is a protein made by cells in the prostate gland (both normal cells and cancer cells) Population: Baseline PSA was calculated for patients whom completed and were used in final analysis
  nanograms per millilitre (ng/mL)
    number analyzed (Participants) | 12
    (all) | 21.1 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Mean Kinetic Parameters Reflecting Fluorocholine (FCH) Fluorine 18 FCH (F-18) Influx (K1)
Description: The average K1 values of primary tumors will be reported along with the standard deviation
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: K1 (min-1)
Groups:
- Choline PET/MR: 11C-Choline: 370MBq Intravenously 18F-Choline: 3MBq/kg Intravenously
  Choline PET/MR
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
K1 (min-1) | 0.562 (0.201)

2. Primary Outcome: Mean Maximum Kinetic Parameters Reflecting F-18 Influx (K1max)
Description: The K1max values of primary tumors will be reported along with the standard deviation
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: K1 (min-1)
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
K1 (min-1) | 0.753 (0.246)

3. Primary Outcome: Average Standardized Uptake Value (SUVavg)
Description: The SUVavg values of primary tumors will be reported along with the standard deviation. Typically, a standardized uptake value (SUV), a quantity that incorporates the patient's size and the injected dose, that is more than 2.0 is considered to be suggestive of malignancy
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
SUV | 6.10 (1.60)

4. Primary Outcome: Mean of the Standardized Uptake Value (SUVmax)
Description: The SUVmax values of primary tumors will be reported along with the standard deviation. Typically, a standardized uptake value (SUV), a quantity that incorporates the patient's size and the injected dose, that is more than 2.0 is considered to be suggestive of malignancy.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
SUV | 8.40 (2.04)

5. Primary Outcome: Sensitivity of Combined Positron Emission Tomography (PET) and Magnetic Resonance (MR) Imaging
Description: Sensitivity (True Positive Rate, TPR) measures the ability of a 11C- and 18F-Choline PET/MR Imaging for Prostate Cancer to correctly identify patient status as respectively diseased or non-dis- eased and is reported as a percentage ranging from 0 -100 with higher percentages indicating a higher sensitivity to identify the prostate cancer using SUVmax . The sensitivity of the combined PET and MR imaging for prediction of pathologic extraprostatic extension will be reported.
Time Frame: Day 1
Measure: Number; unit: percentage of true positives
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
percentage of true positives | 88

6. Primary Outcome: Specificity of of Combined Positron Emission Tomography (PET) and Magnetic Resonance (MR) Imaging
Description: Specificity (True Negative Rate) measures the ability of a 11C- and 18F-Choline PET/MR Imaging for Prostate Cancer to correctly identify patient status as respectively diseased or non-dis- eased and is reported as a percentage ranging from 0 -100 with higher percentages indicating a higher specificity to identify the prostate cancer using SUVmax. The specificity of the combined PET and MR imaging for prediction of pathologic extraprostatic extension will be reported.
Time Frame: Day 1
Measure: Number; unit: percentage of true negatives
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
percentage of true negatives | 100

7. Primary Outcome: Correlation of K1 of Primary Tumors With K1max
Description: A spearman rank correlation test was performed to test the correlation of K1 with K1max. Spearman's correlation coefficient (ρ) determines the strength and direction of the monotonic relationship between two variables. The Spearman correlation coefficient is reported in values from +1 to -1. A ρ= +1 indicates a perfect association of ranks, a ρ = zero indicates no association between ranks and a ρ = -1 indicates a perfect negative association of ranks. The closer ρ is to zero, the weaker the association between the ranks.
Time Frame: Day 1
Measure: Number; unit: Spearman's correlation coefficient (ρ)
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
Spearman's correlation coefficient (ρ) | 0.86

8. Primary Outcome: Correlation of K1 of Primary Tumors With Average Standardized Uptake Value (SUVavg)
Description: A spearman rank correlation test was performed to test the correlation of K1 with the SUVavg of primary tumors. Spearman's correlation coefficient (ρ) determines the strength and direction of the monotonic relationship between two variables. The Spearman correlation coefficient is reported in values from +1 to -1. A ρ= +1 indicates a perfect association of ranks, a ρ = zero indicates no association between ranks and a ρ = -1 indicates a perfect negative association of ranks. The closer ρ is to zero, the weaker the association between the ranks.
Time Frame: Day 1
Measure: Number; unit: Spearman's correlation coefficient (ρ)
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
Spearman's correlation coefficient (ρ) | 0.76

9. Primary Outcome: Correlation of K1max of Primary Tumors With SUVmax
Description: A spearman rank correlation test was performed to test the correlation of K1max with SUVmax. Spearman's correlation coefficient (ρ) determines the strength and direction of the monotonic relationship between two variables. The Spearman correlation coefficient is reported in values from +1 to -1. A ρ= +1 indicates a perfect association of ranks, a ρ = zero indicates no association between ranks and a ρ = -1 indicates a perfect negative association of ranks. The closer ρ is to zero, the weaker the association between the ranks.
Time Frame: Day 1
Measure: Number; unit: Spearman's correlation coefficient (ρ)
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
Spearman's correlation coefficient (ρ) | 0.65

10. Primary Outcome: Correlation of K1max of Primary Tumors With SUVavg
Description: A spearman rank correlation test was performed to test the correlation of K1max with SUVavg. Spearman's correlation coefficient (ρ) determines the strength and direction of the monotonic relationship between two variables. The Spearman correlation coefficient is reported in values from +1 to -1. A ρ= +1 indicates a perfect association of ranks, a ρ = zero indicates no association between ranks and a ρ = -1 indicates a perfect negative association of ranks. The closer ρ is to zero, the weaker the association between the ranks.
Time Frame: Day 1
Measure: Number; unit: Spearman's correlation coefficient (ρ)
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
Spearman's correlation coefficient (ρ) | 0.60

11. Primary Outcome: Correlation of SUVmax of Primary Tumors With SUVavg
Description: A spearman rank correlation test was performed to test the correlation of SUVmax with SUVavg. Spearman's correlation coefficient (ρ) determines the strength and direction of the monotonic relationship between two variables. The Spearman correlation coefficient is reported in values from +1 to -1. A ρ= +1 indicates a perfect association of ranks, a ρ = zero indicates no association between ranks and a ρ = -1 indicates a perfect negative association of ranks. The closer ρ is to zero, the weaker the association between the ranks.
Time Frame: Day 1
Measure: Number; unit: Spearman's correlation coefficient (ρ)
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
Spearman's correlation coefficient (ρ) | 0.65

12. Secondary Outcome: Correlation of SUVmax of Primary Tumors With Serum Prostate-specific Antigen (PSA) Level
Description: A spearman rank correlation test was performed to test the correlation of SUVmax with a patients baseline PSA. Spearman's correlation coefficient (ρ) determines the strength and direction of the monotonic relationship between two variables. The Spearman correlation coefficient is reported in values from +1 to -1. A ρ= +1 indicates a perfect association of ranks, a ρ = zero indicates no association between ranks and a ρ = -1 indicates a perfect negative association of ranks. The closer ρ is to zero, the weaker the association between the ranks.
Time Frame: Day 1
Measure: Number; unit: Spearman rank correlation coefficient (p
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
Spearman rank correlation coefficient (p | 0.71

13. Secondary Outcome: Correlation of SUVmax of Primary Tumors With Pathological Stage
Description: The system of pathological staging is developed by the American Joint Committee on Cancer (AJCC) and is divided into 5 stages: stage 0 (zero) and stages I through IV (1 through 4). A spearman rank correlation test was performed to test the correlation of SUVmax with a patient's baseline pathological stage. Spearman's correlation coefficient (ρ) determines the strength and direction of the monotonic relationship between two variables. The Spearman correlation coefficient is reported in values from +1 to -1. A ρ= +1 indicates a perfect association of ranks, a ρ = zero indicates no association between ranks and a ρ = -1 indicates a perfect negative association of ranks. The closer ρ is to zero, the weaker the association between the ranks.
Time Frame: Day 1
Measure: Number; unit: Spearman rank correlation coefficient (p
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
Spearman rank correlation coefficient (p | 0.59

14. Secondary Outcome: Correlation of SUVmax of Primary Tumors With Post-surgical Cancer of the Prostate Risk Assessment (CAPRA) Scores
Description: The CAPRA is a 5 item questionnaire completed by the clinicians with a total score range from 0-10 calculated using points assigned to: age at diagnosis, PSA at diagnosis, Gleason score of the biopsy, clinical stage and percent of biopsy cores involved with cancer. A CAPRA score of 0 to 2 indicates low-risk, a score of 3 to 5 indicates intermediate-risk, and a score of 6 to 10 indicates high-risk. A spearman rank correlation test was performed to test the correlation of SUVmax with a patient's CAPRA score after surgery. Spearman's correlation coefficient (ρ) determines the strength and direction of the monotonic relationship between two variables. The Spearman correlation coefficient is reported in values from +1 to -1. A ρ= +1 indicates a perfect association of ranks, a ρ = zero indicates no association between ranks and a ρ = -1 indicates a perfect negative association of ranks. The closer ρ is to zero, the weaker the association between the ranks.
Time Frame: After surgery, Up to 6 months
Measure: Number; unit: Spearman rank correlation coefficient (p
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
Spearman rank correlation coefficient (p | 0.72

15. Secondary Outcome: Comparison of SUVmax of Primary Tumors With Post-surgical Cancer of the Prostate Risk Assessment (CAPRA) Score Groups
Description: The CAPRA is a 5 item questionnaire completed by the clinicians with a total score range from 0-10 calculated using points assigned to: age at diagnosis, PSA at diagnosis, Gleason score of the biopsy, clinical stage and percent of biopsy cores involved with cancer. A CAPRA score of 0 to 2 indicates low-risk, a score of 3 to 5 indicates intermediate-risk, and a score of 6 to 10 indicates high-risk. A Mann-Whitney U test was performed to compare the SUVmax with patients classified as intermediate-risk and high risk based on their CAPRA Score. Means and standard deviations will be reported.
Time Frame: After surgery, Up to 6 months
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | Choline PET/MR
Number analyzed (Participants) | 12
SUVmax
  Intermediate Risk Group | 9.53 (1.48)
  High Risk Group | 6.24 (1.26)
Statistical Analysis 1: Comparison: Choline PET/MR; Test type: Other; p < .008, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 day, up to 30 minutes after injection
Description: Only NCI Common Terminology Criteria for Adverse Events (CTCAE) of grade 3 or higher were collected for this study.
Arm/Group | Diagnostic 11C- and 18F-choline PET/MR Imaging
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes